CLINICAL TRIAL: NCT00665301
Title: Validation Study Comparing the Cardiac Output Pulmonary Arterial Catheter (Swan Ganz) to the FloWave™ 1000 Device
Brief Title: Cardiac Output Pulmonary Arterial Catheter Compared to FloWave™ 1000
Status: Completed | Type: Observational
Sponsor: Woolsthorpe Technologies, LLC (Industry)
Responsible Party: Jeannie Brooks, RN, BSN/Director, Clinical Trials, Woolsthorpe Technologies, LLC
Other Study IDs: WFW-019
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Congestive Heart Failure; Ischemic Cardiomyopathy; Mitral Valve Prolapse; Mitral Regurgitation; Aortic Valve Disease; Tricuspid Regurgitation
Keywords: Non-invasive Cardiac Output
MeSH Terms: conditions — Heart Failure; Mitral Valve Prolapse; Mitral Valve Insufficiency; Aortic Valve Disease; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare cardiac output results obtained using the thermodilution push technique with the Pulmonary Arterial Catheter (PAC) to the predicted cardiac output results obtained from the non-invasive FloWave™ 1000 device.

ELIGIBILITY:
Inclusion Criteria:

* Adults Only: The FloWave device is intended for use on adult patients only. All subjects will be 18 years or older.
* Existing placement of a Pulmonary Arterial Catheter placed for medical reasons other than our study.

Exclusion Criteria:

* Patients with aortic balloon pumps and cardiac mechanical assist devices will be excluded from study enrollment if the devices are present during the screening process. If patients have cardiac assist devices inserted after enrollment in the study, cardiac output data will be collected with both the PAC and FloWave device and will be evaluated as a subset analysis population at the conclusion of the study.
* Patients with intracardiac shunts will be excluded from this study.
* FloWave cardiac output determinations are dependent on detection of a pulse. If no peripheral pulse can be detected the device will not be able to perform a measurement and this will be indicated to the user.
* Patients who are not in a steady hemodynamic state shall be excluded from the study.
* Presence of arrhythmias: Patients with arrhythmias are excluded from the study when not in a steady hemodynamic state. If a patient has a history of arrhythmia or is currently experiencing an arrhythmia but is in a maintained hemodynamic state, they will not be excluded from enrollment into the study. Their clinical symptoms and cardiac rhythm will be evaluated and noted in the patient data record.
* Inability or unwillingness of subject or the subject's legally authorized representative to give informed consent.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient that has a Swan Ganz PAC catheter in place.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Correlation of FloWave 1000™ Device estimated cardiac output results with Pulmonary Catheter Themodilution Push derived cardiac output results. | Simultaneous data collection during procedure. No follow-up required.

CONTACTS AND LOCATIONS:
Overall Officials: Jim M. Perry, M.D., Study Director
Locations (3):
- United States (3):
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Hospital, Nashville, Tennessee
  - Texas Heart Institute - St. Luke's Hospital, Houston, Texas

REFERENCES:
- See also: Click here for more information about this study: Cardiac Output Pulmonary Arterial Catheter Compared to FloWave™ 1000 — http://www.woolsthorpe.com